CLINICAL TRIAL: NCT04553276
Title: Co-morbidity and Refractory Asthma - UK Severe Asthma Registry
Acronym: UKSAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University, Belfast (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); University Hospitals, Leicester (Other); Nottingham University Hospitals NHS Trust (Other); University Hospitals of North Midlands NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); The Leeds Teaching Hospitals NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); Oxford University Hospitals NHS Trust (Other); University Hospital Plymouth NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other); Taunton and Somerset Hospital (Other); Lancashire Teaching Hospitals NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Liam Heaney, Professor of Respiratory Medicine, Queen's University, Belfast
Other Study IDs: DB/SAR2020
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A "Clinical Registry" is a database which contains clinical information about people with different medical conditions. They are used in many countries throughout the world to help medical teams to better understand specific diseases and improve the care and treatment of patients.

The UK Severe Asthma Registry has been collecting data on patients attending Severe Asthma Clinics in the UK since 2007.

After obtaining appropriate consent from patients to use their information, data is entered by the patient's own clinical team and it is kept up-to-date to follow clinical progress and response to treatments. Very strict controls are in place to make sure individuals cannot be identified from the Registry and all information available from the National Registry is anonymous.

Apart from the local clinic team, occasionally trusted third parties will also be able to identify you, if required to do so, on a strict need-to-know basis. This is necessary to ensure that the Registry works efficiently, or as a part of a Research Project, previously approved by a Research Ethics Committee.

Data from the Registry has a number of uses including judging which severe asthma treatments are of greater benefit, to identify different subgroups of severe asthma and trial new therapies and to provide information for planning future services for people with severe asthma. The use of any information from the UK Severe Asthma Registry requires approval of the Steering Committee which is made up of the refractory asthma specialists from across the UK and who will have access to data protection, legal and ethics expertise where necessary, to safeguard the use of data.

If the Registry closes, data will be returned to the local clinic team if requested, otherwise it will be destroyed. Participation is entirely voluntary and patients can withdraw consent form the Registry at any time by informing their local clinical team. The Data Controller from the UK Severe Asthma Registry is Queen's University Belfast and the Data Processor is Dendrite Clinical Services Ltd which is a commercial provider of database and registry systems.

DETAILED DESCRIPTION:
There are currently 14 Networks of UK dedicated Specialist Difficult Asthma Services submitting data to the UK Registry: Belfast City Hospital; Royal Brompton & Harefield, London; Birmingham Regional Severe Asthma Service; South Thames & Kent Severe Asthma Service; East Midlands Severe Asthma Network; North West Midlands Severe Asthma Service; Yorkshire Asthma MDT; East of England Severe Asthma Network; Wessex Severe Asthma Network; South West Asthma Network; North West Asthma Network, Newcastle Severe Asthma Network and Greater Glasgow & Clyde.

The Registry was set up to standardise clinical services in the UK and facilitate research into patients with difficult asthma. Patients that attend difficult asthma services across the UK are approached to give consent for inclusion. The Registry is hosted online by Dendrite Clinical Systems and admits password protected anonymised data, after fully informed written consent is obtained from patients (see Patient Information and Consent sheets). The individual centre data can be downloaded locally by registered users for audit purposes. The Registry records patient demographics including gender, age at diagnosis, race, occupation, smoking status, BMI. Disease characteristics such as asthma medication, unscheduled healthcare visits, exacerbations, hospital and ICU admissions, blood and sputum investigations, allergen testing, pulmonary function are also recorded in the registry.

Subjects have been entered into the Registry in a non-selected manner and there are currently over 4800 subjects in the Registry with detailed demographic, disease characteristics and health outcome data. Of these subjects, the majority after detailed assessment fulfil the American Thoracic Society definition of refractory asthma, whilst others after detailed assessment are identified as having non-refractory asthma.

The Registry has also been expanded to collect data on bronchial thermoplasty in line with NICE Guidance on bronchial thermoplasty for severe asthma (http://www.nice.org.uk/guidance/ipg419).

the Registry with detailed demographic, disease characteristics and health outcome data.

As part of NHS England Central Commissioning for Specialist Severe Asthma Services, all specialist centres in the UK will be required to input data into the Registry to enable benchmarking between centres.

ELIGIBILITY:
Inclusion Criteria:

1. Referral to a specialist severe asthma clinic in the UK due to inadequate asthma control

Exclusion Criteria: None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that are referred to specialist severe asthma services across the UK. The majority of patients after detailed assessment fulfill the American Thoracic Society definition of refractory asthma, whilst others after detailed assessment are identified as having non-refractory asthma.
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2025-08-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with no systemic corticosteroid exposure in most recent 12 month follow-up period | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UK SAR Database with list of active projects — https://hscn.e-dendrite.com/csp/asthma/frontpages/Registry-projects.pdf